CLINICAL TRIAL: NCT05923021
Title: A Randomized Controlled Study on the Treatment of Moderate Depressive Disorder With Cheek Acupuncture
Brief Title: Moderate Depressive Disorder With Cheek Acupuncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-KLS-049-01
Record Dates: First submitted 2023-05-19; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Acupuncture; Depression
Keywords: cheek acupuncture; depression; MDD; RCT research; functional links
MeSH Terms: conditions — Depression | interventions — Sertraline

STUDY DESIGN:
Intervention Model Description: The specific method is to randomly assign 126 patients with moderate depressive disorder to cheek acupuncture group, sham cheek acupuncture group and drug group, evaluate the treatment effect with HAMD-17, PSQI and HAMA, observe the improvement of cheek acupuncture on depression, anxiety and sleep of patients with moderate depressive disorder, and observe the changes of functional links in various brain regions of patients in each group before and after treatment through resting state functional magnetic resonance imaging technology.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The project adopts a central random system for random grouping and obtains a random number. The random number does not reflect grouping information, so blind method can be implemented for subjects and evaluators. However, due to the setting of sham cheek acupuncture in the project grouping, blind method can't be implemented for researchers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cheek acupuncture treatment group (Experimental): Needle selection: Select disposable trocars（φ0.18 × 25mm） (Wujiang Jiachen acupuncture and moxibustion Instrument Co., Ltd.) .
  Acupoints selection: bilateral Sanjiao points, bilateral head points, bilateral neck points, Needling depth: about 5mm-7.5mm, Needle retaining time: 30 minutes, course of treatment: 3 times a week, with a total of 36 cheek acupuncture treatments for 12 weeks.
  Interventions: Other: cheek acupuncture
- Sham cheek acupuncture treatment group (Sham Comparator): Needle selection: Select disposable flat head trocars（φ0.18 × 25mm） (Wujiang Jiachen acupuncture and moxibustion Instrument Co., Ltd.) .
  Acupoints selection: Translate the bilateral Sanjiao points forward by 1cm（towards the front midline of the body）, translate the bilateral head points forward by 1cm, bilateral back points, Needling depth: Retained on the surface of the skin with the help of a cannula， Needle retaining time: 30 minutes, course of treatment: 3 times a week, with a total of 36 times of cheek acupuncture treatments for 12 weeks.
  Interventions: Other: cheek acupuncture
- Drug group (Active Comparator): Drug name: Sertraline Hydrochloride Tablets (trade name: Levofloxacin Sertraline, produced by Pfizer Pharmaceutical Co., Ltd., batch number: H10980141),
  Dosage form: tablets
  Usage: Take orally. 50 mg/d, taken after breakfast.
  Depending on the patient's condition, the dosage can be increased to 200mg/d, taken after breakfast, or divided twice a day after meals
  Treatment cycle: a total of 12 weeks.
  Interventions: Other: cheek acupuncture

INTERVENTIONS:
Other: cheek acupuncture — Cheek acupuncture therapy refers to a new painless acupuncture therapy for treating systemic diseases by acupuncture at specific points on the cheek. This therapy was founded by Professor Wang Yongzhou, a scholar in France. Cheek acupuncture therapy takes the Yellow Emperor's Internal Classic as the theoretical basis, and organically integrates holographic theory, the theory of ascending and descending qi, the theory of Big Three Jiao, the theory of simultaneous treatment of mind and body, and the theory of the book of Changes.In this study, we use the big three jiao points, head points, and neck points in cheek acupuncture therapy to treat depression. These acupoints are considered effective in long-term clinical applications.
  Other Names: Sertraline Hydrochloride Tablets

SUMMARY:
This study intends to use a randomized controlled clinical study to clarify the clinical efficacy of cheek acupuncture therapy in patients with moderate depressive disorder. And also to find the antidepressant mechanism of cheek acupuncture therapy on moderate depressive disorder by using resting state functional magnetic resonance imaging. The specific method is to randomly assign 126 patients with moderate depressive disorder to cheek acupuncture group, sham cheek acupuncture group and drug group, evaluate the treatment effect with HAMD-17, PSQI and HAMA, observe the improvement of cheek acupuncture on depression, anxiety and sleep quality of patients with moderate depressive disorder, and observe the changes of functional links in various brain regions of patients in each group before and after treatment through resting state functional magnetic resonance imaging technology.

DETAILED DESCRIPTION:
Cheek acupuncture therapy refers to a new painless acupuncture therapy for treating systemic diseases by acupuncture at specific points on the cheek. This therapy was founded by Professor Wang Yongzhou, a scholar in France. Cheek acupuncture therapy takes the Yellow Emperor's Internal Classic as the theoretical basis, and organically integrates holographic theory, the theory of ascending and descending qi, the theory of Big Three Jiao, the theory of simultaneous treatment of mind and body, and the theory of the book of Changes. After long-term and extensive clinical practice and continuous experience summary, a relatively independent and complete treatment system has been formed. Since its initial discovery in 1991, cheek acupuncture has undergone clinical observation and verification by numerous doctors for nearly 100000 times. Its therapeutic effect is stable and reliable, and it has a strong therapeutic advantage for psychosomatic diseases represented by depression. The members of the research group have been learning about cheek acupuncture since 2017 and have applied it to the treatment of patients with depression, achieving satisfactory clinical efficacy.

Major depressive disorder (MDD) is a type of disorder with high incidence, recurrence, disability, and the risk of suicide for severe mental disorders with a high suicide rate is about 20 times higher than that of the general population. The main clinical features of this disease are low mood, decreased interest, and lacking in strength. Many patients also experience symptoms such as cognitive decline, autonomic dysfunction, sleep disorders, and altered appetite. A 2013 study on the global burden of disease pointed out that depression is the second largest burden disease worldwide, with a prevalence rate of 6.7% in China About 9%, with a total number of approximately 95 million cases. Deeply exploring the pathogenesis of depression and exploring new antidepressant therapies have significant practical significance.

In this situation, the investigators design a randomized controlled clinical study, firstly to clarify the cure effect of cheek acupuncture therapy, secondly to find the central mechanism of it on antidepressant effect.The specific method is to randomly assign 126 patients with moderate depressive disorder to cheek acupuncture group, sham cheek acupuncture group and drug group, evaluate the treatment effect with HAMD-17, PSQI and HAMA, observe the improvement of cheek acupuncture on depression, anxiety and sleep of patients with moderate depressive disorder, and observe the changes of functional links in various brain regions of patients in each group before and after treatment through resting state functional magnetic resonance imaging technology.

ELIGIBILITY:
Inclusion Criteria:

* ① Conforming to the diagnostic standards of traditional Chinese and Western medicine;

  * Age range from 10 to 65 years old;

    * HAMD-17 scores>14 ;

      * Sign an informed consent form (Minors need to obtain recognition from their guardians and have their informed consent signed by their guardians) and voluntarily participate in this study.

Only those who meet the above 4 criteria can be included in the study.

Exclusion Criteria:

* ①Individuals with significant suicidal tendencies;

  * Previously diagnosed with intellectual disabilities, schizophrenia, bipolar disorder, substance abuse (such as alcohol dependence), or other mental disorders;

    * Epilepsy history or strong positive epilepsy family history, brain organic disease and serious physical disease history;

      * Individuals who are taking antidepressants within 6 weeks (including 6 weeks);

        * Pregnancy, preparation or lactation period;

          * Patients with skin lesions or skin diseases, severe diabetes, tumors and dysfunction of important organs, or severe internal diseases such as liver, kidney, cardiovascular, endocrine, respiratory and hematopoietic systems;

            ⑦ Contraindications for fMRI examination, such as pacemakers, cardiac stents, and claustrophobia;
            * Patients with other central or peripheral neuropathy.

Those who meet any of the above criteria will be excluded from the study

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change HAMD-17 score is being assessed at different time points | Baseline, 1week, 2 weeks, 3weeks, 4weeks, 8weeks, 12 weeks,20 weeks
  The most commonly used scale for clinical assessment with depression. A score more than or equal to 24 indicates severe depression, a score more than or equal to 17 and less than 24 indicates moderate depression, and a score less than 7 indicates no depression.

SECONDARY OUTCOMES:
Change PSQI score is being assessed at different time points | Baseline, 1week, 2 weeks, 3weeks, 4weeks, 8weeks, 12 weeks,20 weeks
  It will be used to evaluate the sleep quality of subjects in the past month, the scale consists of 18 self-assessment items combined into 7 factors, each factor scored on a 0-3 scale, and the total score of each factor is the PSQI total score. The higher the score, the poorer the sleep quality. Generally, a score of 7 is the cutoff value, while a PSQI ≥ 8 indicates poor sleep quality.
Change HAMA score is being assessed at different time points | Baseline, 1week, 2 weeks, 3weeks, 4weeks, 8weeks, 12 weeks,20 weeks
  It is an anxiety assessment scale with a total of 14 items, and each symptom is divided into 0-4 points. A score less than 7 indicates no anxiety, more than or equal to 7 indicates possible anxiety.

IPD SHARING:
Plan to Share IPD: No